CLINICAL TRIAL: NCT01470391
Title: "A Comparison of the Efficacy of the Adductor-Canal-Blockade Versus the Femoral Nerve Block on Muscle Strength, Pain and Mobilization After Total Knee Arthroplasty: a Randomized Study
Brief Title: Adductor-Canal-Blockade Versus the Femoral Nerve Block Effect on Muscle Strength, Pain and Mobilization After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-PJ-11
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Total Knee Arthroplasty
Keywords: Adductor-Canal-Blockade; Femoral Nerve Block; Postoperative Pain; Total Knee Arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adductor-Canal-Blockade (Experimental)
  Interventions: Procedure: Adductor-Canal-Blockade
- Femoral Nerve Block (Active Comparator)
  Interventions: Procedure: Femoral Nerve Block

INTERVENTIONS:
Procedure: Adductor-Canal-Blockade — US-guided Adductor-Canal-Blockade with Ropivacaine
  Arms: Adductor-Canal-Blockade
Procedure: Femoral Nerve Block — US-guided Femoral Nerve Block with Ropivacaine
  Arms: Femoral Nerve Block

SUMMARY:
The aim of this study is to investigate the efficacy of the Adductor-Canal-Blockade versus the Femoral Nerve Block on muscle strength, pain and mobilization after total knee arthroplasty. We hypothesize that the Adductor-Canal-Blockade has the same effect on pain and morphine consumption as the Femoral Nerve Block, but without the same reduction in quadriceps muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* BMI > 18 og < 40
* total knee arthroplasty in spinal anesthesia

Exclusion Criteria:

* Can not cooperate to the exam
* Do not speak or understand Danish
* Drug allergy
* Alcohol or drug abuse
* Daily consumption of strong opioids
* Rheumatoid arthritis
* Intake of glucocorticoids
* Effect of spinal anesthesia stopped prior to performing the regional block

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The difference in quadriceps muscle strength between the Adductor-Canal-Blockade and the femoral nerve block | 24 h postoperatively

SECONDARY OUTCOMES:
The difference in adductor muscle strength between the Adductor-Canal-Blockade and the Femoral Nerve Block | 24 h postoperatively
Pain during flexion of the knee | 2-24 hours
  0-100 mm at a visual analogue scale (VAS), calculated as the area under the curve for the interval 2-24 hours postoperatively.
Pain at rest | 2-24 hours
  0-100 mm at a visual analogue scale (VAS), calculated as the area under the curve for the interval 2-24 hours postoperatively.
Total morphine consumption | 0-24 hours
Postoperative nausea | 2-24 hours
Postoperative vomiting | 0-24 hours
Sedation | 2-24 hours
Zofran consumption | 0-24 hours
  Number of patients recieveing zofran postoperatively
The difference in mobilization between the groups | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Anaesthesia, Copenhagen University Hospital, Frederiksberg, Frederiksberg, Frederiksberg, Denmark

REFERENCES:
- [Derived] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608